CLINICAL TRIAL: NCT05198115
Title: Premenstrual Syndrome in Young Women With Eight Weeks of Aerobic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Said Ali, dr ahmedsaidali MCs candidate Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3574
Record Dates: First submitted 2021-12-19; First posted 2022-01-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Aerobic Exercise; Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Eight Weeks of Aerobic Exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic group (Active Comparator): The intervention consisted of aerobic exercise training, which was taught to participants face-to-face at a meeting. At the end of the session, we provided the intervention group with CDs and educational posters containing all the exercises
  Interventions: Behavioral: aerobic exercise
- Eight Weeks of Aerobic Exercise (Placebo Comparator): The control group was subjected to all the pre-and post-assessments but were not asked to perform the exercise intervention. Instead, we phone-called them to give a reminder for filling out the questionnaires.
  Interventions: Behavioral: aerobic exercise

INTERVENTIONS:
Behavioral: aerobic exercise — aerobic training for 8 weeks, 3 times a week, and 60 min each time

SUMMARY:
The premenstrual syndrome includes physical and psychological symptoms that occur at the end menstrual cycle and exercise is one of the ways to reduce symptoms. The aim of this study was to determine the effect of a regular 8-week aerobic exercise program on psychological symptoms of premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome is characterized by the presence of both physical and behavioral (including affective) symptoms that occur repetitively in the second half of the menstrual cycle and interfere with some aspects of the woman's life(1). The core symptoms of PMS include affective symptoms, such as irritability, depression, anxiety, and somatic symptoms, such as breast pain, bloating, swelling, and headache (2). Women with moderate to severe PMS symptoms had a reduction in health-related quality of life(3) and work productivity, increased work absenteeism, and visits to ambulatory healthcare providers (4), so the treatment of this syndrome is essential.

ELIGIBILITY:
Inclusion Criteria:

* young women aged 18-25 years with a body mass index (BMI): 18-25 kg/m2, having regular menstrual cycles of 23-35 days duration, no previous practice of aerobic exercise, free from musculoskeletal injury, not using oral contraceptive pills or taking any psychotropic agents, having no depression or genital tract diseases

Exclusion Criteria:

* pregnancy, contraindications to physical exercise, metabolic or cardiorespiratory illness, cigarette smokers, women who recover from a major injury or using anti-inflammatory, hyperlipidemia or hypertension medications, any abnormality in ovulation, and women with diabetes mellitus, thyroid, pituitary, or ovarian disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pms only for women
Enrollment: 50 (Estimated)
Dates: Start 2022-02-25 (Estimated); Primary Completion 2022-04-25 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Emotional (EM) scale | eight weeks
  emotional scale from [0 to 10]

IPD SHARING:
Plan to Share IPD: No